CLINICAL TRIAL: NCT01714908
Title: A Multicenter, Randomized, Open-label, Phase II Study to Evaluate the Efficacy and Safety of Erlotinib Versus Etoposide Plus Cisplatin With Concurrent Radiotherapy in Unresectable Stage III Non-small Cell Lung Cancer (NSCLC) With Activating Mutation of Epidermal Growth Factor Receptor (EGFR) in Exon 19 or 21
Brief Title: Phase II Study of Erlotinib With Concurrent Radiotherapy in Unresectable NSCLC With Activating Mutation of EGFR in Exon 19 or 21
Acronym: RECEL
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jinming Yu (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor-Investigator, Jinming Yu, Professor, Shandong Cancer Hospital and Institute
Organization: Shandong Cancer Hospital and Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ML28545
Record Dates: First submitted 2012-10-23; First posted 2012-10-26 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; EGFR mutation; unresectable; erlotinib; concurrent radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erlotinib w Concurrent Radiotherapy (Experimental): erlotinib 150mg oral daily up to 2 years concurrent radiotherapy total dose 60-66 Gray (Gy) in 2 Gray (Gy) fractions. One fraction per day, and 5 fractions per week.
  Interventions: Other: Erlotinib w Concurrent Radiotherapy
- etoposide/cis-platin (EP) w Concurrent Radiotherapy (Active Comparator): etoposide 50mg/m2 on D1-5 and D29-33 cis-platin 50mg/m2 on D1, D8, D29 and D36 concurrent radiotherapy total 60-66 Gray (Gy) in 2 Gray (Gy) fractions. One fraction per day, 5 fractions per week.
  Interventions: Other: etoposide/cis-platin (EP) w Concurrent Radiotherapy

INTERVENTIONS:
Other: Erlotinib w Concurrent Radiotherapy
  Arms: Erlotinib w Concurrent Radiotherapy
Other: etoposide/cis-platin (EP) w Concurrent Radiotherapy — Etoposide / Cis-platin w Concurrent Radiotherapy
  Arms: etoposide/cis-platin (EP) w Concurrent Radiotherapy

SUMMARY:
Erlotinib with concurrent radiotherapy has superior efficacy and comparable safety profile in unresectable stage III non-small cell lung cancer (NSCLC) patients with activating mutation of epidermal growth factor receptor (EGFR) in exon 19 or 21 versus etoposide plus cis-platin with concurrent radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC confirmed by histopathology or cytology;
* Stage IIA or IIIB NSCLC according to Tumor Node Metastasis (TMN) staging of Lung Staging Standard version 7 2009, and be unresectable;
* Has active mutation of EGFR in exon 19 or 21;
* Has measurable lesion [according to Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, must have at least one evaluable lesion with the longest dimension >= 10mm; if the evaluable lesion is lymph node, the shortest dimension should be measured and >=15mm];
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-1;
* expectancy life >= 12 weeks;

Exclusion Criteria:

* Had be treated by HER-targeting agents;
* Had systemic anit-NSCLC treatments;
* Had local radiotherapy for NSCLC;
* Has upper gastrointestinal physiological disorders, or malabsorption syndrome, or intolerance of oral medication, or active peptic ulcer;
* Diagnosed other malignant tumor besides NSCLC within 5 years prior the study treatment (except having simple surgical resection with 5-year disease free survival, cured in situ of cervical carcinoma, cured basal cell carcinoma and bladder epithelial tumor);
* Any evidence to indicate moderate or severe chronic obstructive pulmonary disease (COPD);
* Known hypersensitivity to platinum, etoposide, EGFR-Tyrosine Kinase Inhibitor (TKI) agents or relevant components in the formulation;
* Uncontrolled eye inflammation or infection, or any potential circumstances lead to eye inflammation or infection;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2012-12-14 (Actual); Primary Completion 2018-08-20 (Estimated); Study Completion 2018-10-20 (Estimated)

PRIMARY OUTCOMES:
Progress Free Survival (PFS) | 5 years
  The time frame from the randomization to the first confirmed disease progression or any cause to death (dependent on which comes first)

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute; Shenglin Ma, PhD, Principal Investigator — The First People's Hospital of Hangzhou; Conghua Xie, PhD, Principal Investigator — Zhongnan Hospital; Ming Chen, PhD, Principal Investigator — Zhejiang Cancer Hospital; Gang Wu, PhD, Principal Investigator — Tongji Medical College, Huazhong University of Science and Technology, Wuhan Union Hospital; Jianhua Wang, PhD, Principal Investigator — Henan Cancer Hospital; Jiancheng Li, PhD, Principal Investigator — Fujian Province Cancer Hospital; Zhengfei Zhu, PhD, Principal Investigator — Fudan University; You Lu, PhD, Principal Investigator — West China Hospital, West China School of Medicine, Sichuan University; Lvhua Wang, PhD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Guangying Zhu, PhD, Principal Investigator — Peking University Cancer Hospital & Institute; Tingyi Xia, PhD, Principal Investigator — Chinese PLA General Hospital; Chun Han, PhD, Principal Investigator — Hebei Medical University Fourth Hospital; Guang Li, PhD, Principal Investigator — First Hospital of China Medical University; Zhiyong Yuan, PhD, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital; Qin Lin, PhD, Principal Investigator — The First Affiliated Hospital of Xiamen University; Qibin Song, PhD, Principal Investigator — Renmin Hospital of Wuhan University; Yaping Xu, PhD, Principal Investigator — Zhejiang Cancer Hospital; Bing Lu, PhD, Principal Investigator — Cancer Hospital of Guizhou Province; Baolin Qu, PhD, Principal Investigator — Chinese PLA General Hospital
Locations (19):
- China (19):
  - Cancer Institute & Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - The General Hospital of the People's Liberation Army, Beijing, Beijing Municipality
  - Fujian Province Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - Guizhou Cancer Hospital, Guiyang, Guizhou
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Wuhan Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - Renmin Hospital of Wuhan University, Wuhan, Hubei
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Cancer Hospital and Institute, Jinan, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital, West China School of Medicine, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - The First People's Hospital of Hangzhou, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang